CLINICAL TRIAL: NCT05567133
Title: Development of Clinical Prediction Models for Pulmonary Outcomes in Sarcoidosis
Brief Title: Risk Indicators of Sarcoidosis Evolution-Unified Protocol
Acronym: RISE-UP
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Vanderbilt University Medical Center (Other); University of Texas, Southwestern Medical Center at Dallas (Other); Wayne State University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: P0551258; R01HL157533 (NIH)
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: sarcoid, lung, immune
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — blood samples for serum isolation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop prediction models that can prognosticate patients with sarcoidosis using clinical data and blood markers that can be obtained during a clinic visit.

DETAILED DESCRIPTION:
The purpose of this study is to develop prediction models that can prognosticate patients with sarcoidosis using clinical data and biological markers that can be obtained during a clinic visit.

Primary Aim/Objective The primary objective of this study is to determine which clinical features measured during a routine clinic visit are risk factors for progression of pulmonary sarcoidosis over the follow-up period in adults with pulmonary sarcoidosis.

Secondary Aim/Objectives The secondary objective is to determine if blood biomarkers measured during a routine clinic visit can improve the risk assessment for progression of pulmonary sarcoidosis over the follow-up period.

The investigators will measure two types of blood markers to achieve this goal:

* Clinically available blood markers that are available in most clinical labs
* Blood proteins and gene expression that reflect interferon inflammation and are not currently available as tests in clinical labs

ELIGIBILITY:
Inclusion Criteria:

1. Adults with a diagnosis of sarcoidosis over the age of 18
2. Case definition: we will follow the 1999 statement on sarcoidosis published by the American Thoracic Society for diagnosis which includes tissue biopsy confirmation and exclusion of alternative diagnoses including beryllium sensitization/chronic beryllium disease, mycobacterial, viral, and/or fungal infection

Exclusion Criteria:

1. Inability to tolerate study procedures as determined by the investigator
2. Pregnant or breastfeeding
3. Concurrent medical diagnoses that would influence the expression of biomarkers will be considered an exclusion criterion. This includes diseases such as common variable immunodeficiency, HIV infection, or autoimmune diseases
4. Concurrent interstitial lung diseases such as hypersensitivity pneumonitis or idiopathic pulmonary fibrosis
5. Hematocrit (Packed Cell Volume) < 25%

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adults who meet criteria for the diagnosis of pulmonary sarcoidosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2030-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Forced Vital Capacity in Liters | Baseline and 24 months
  Forced vital capacity (FVC) is the total amount of air in liters exhaled during a forced maneuver.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Koth, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drake WP, Hsia C, Samavati L, Yu M, Cardenas J, Gianella FG, Boscardin J, Koth LL. Risk Indicators of Sarcoidosis Evolution-Unified Protocol (RISE-UP): protocol for a multi-centre, longitudinal, observational study to identify clinical features that are predictive of sarcoidosis progression. BMJ Open. 2023 Apr 3;13(4):e071607. doi: 10.1136/bmjopen-2023-071607. PMID 37012011